CLINICAL TRIAL: NCT03236324
Title: Efficacy of Ultrasound-guided Transversalis Fascia Plane Blocks for Post-cesarean Section Analgesia: a Randomized Double Blinded Control Study
Brief Title: Transversalis Fascia Plane Blocks for Analgesia Post-cesarean Delivery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB15-2238
Record Dates: First submitted 2017-07-25; First posted 2017-08-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cesarean Delivery
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TFP block with saline (Placebo Comparator): Placebo bilateral ultrasound-guided nerve block [transversalis fascia plane (TFP) block] with 40 mL saline, single shot
  Interventions: Device: ultrasound-guided nerve block; Drug: Saline
- TFP block with local anesthetic (Experimental): Experimental bilateral ultrasound-guided nerve block [transversalis fascia plane (TFP) block] with local anesthesic of Bupivacaine-epinephrine [0.25% bupivacaine with 2.5 mcg/mL epinephrine 40 mL (maximum 2.5 mg/kg)], single shot
  Interventions: Device: ultrasound-guided nerve block; Drug: Bupivacaine-epinephrine

INTERVENTIONS:
Device: ultrasound-guided nerve block — Transversalis fascia plane (TFP) block, ultrasound-guided
Drug: Saline — 20 mL 0.9% saline administered on each side as bilateral TFP blocks
  Arms: TFP block with saline
Drug: Bupivacaine-epinephrine — 20 mL bupivacaine 0.25% with epinephrine 2.5 mcg/mL to a maximum of 2.5mg/kg administered on each side as bilateral TFP blocks
  Arms: TFP block with local anesthetic

SUMMARY:
The aim of this study is to assess the efficacy of a bilateral TFP block in parturients undergoing cesarean delivery (CD) by evaluating postoperative opioid consumption and numeric rated pain scores in two groups (TFP block with saline (control) and TFP block with local anesthetic (treatment)). Women (American Society of Anesthesiologists physical status Class 1-3) at term gestation with singleton pregnancies undergoing an elective CD under spinal anesthesia at the South Health Campus will be consented to participate in the study. Patients will be randomly assigned using a computer-generated table of random numbers to two groups. Group allocations will be concealed. All patients will receive spinal anesthesia with spinal Morphine according to our institutional protocol. At the end of surgery, randomized patients will receive either ultrasound-guided bilateral TFP blocks with 0.25% bupivacaine with 2.5 mcg/ml epinephrine 40 ml total or maximum 2.5 mg/kg (Group 1) or 40 mL saline (Group 2) by 2 anesthesiologists experienced in performing this block.

DETAILED DESCRIPTION:
Caesarean delivery (CD) is one of the most commonly performed surgical procedures with an estimated annual frequency of 27% in Alberta between 2007-2011. Poorly controlled postsurgical pain is associated with an increase in morbidity. Untreated or undertreated pain can lead to respiratory infections secondary to splinting and shallow breathing. Excessive pain also reduces and delays ambulation, which can lead to both an increase in the incidence of deep vein thrombosis (DVT) and delay recovery and readiness for discharge. Poorly controlled pain may also lead to the development of chronic postsurgical pain. The optimal form of postoperative analgesia following CD is not known. Most postoperative analgesic protocols for CD, despite being multimodal in nature, rely heavily on opioid medications both orally and intrathecally for analgesia. These medications, however, are not without serious side effects such as nausea, vomiting, sedation, addiction or dependence, and respiratory depression as well as expression in breast milk which may put infants at risk of side effects as well. Thus, an effective alternative analgesic modality analgesia in these patients which produces both improved pain control and reduced side effects is desired. The TFP block represents a promising alternative, which may fulfill this role in complementing multimodal analgesia for patients undergoing CD and reducing opioid administration.

This project aims to elucidate information regarding alternative interventions for postoperative analgesia following CD. While the most common analgesic regimen of intrathecal and oral opioids, acetaminophen, and NSAIDS for postoperative analgesia is effective, it is not appropriate for all patients. For those who cannot receive intrathecal opioids (e.g. those with allergies to opioid medications, or those who are undergoing CD under general anesthetic), alternative analgesic modalities are important to provide adequate multimodal analgesia and minimize side effects of each of the analgesic medications. Additionally, this aforementioned common analgesic pathway may itself be further optimized through the addition of new analgesic techniques. The Transversalis Fascia Plane (TFP) block is a nerve block, which could potentially target nerves responsible for transmitting pain following CD, and represents a promising novel analgesic modality.

ELIGIBILITY:
Inclusion Criteria:

* elective Cesarean delivery with spinal anesthesia at South Health Campus
* term gestation with a singleton pregnancy
* American Society of Anesthesiologists' (ASA) physical status Class 1-3

Exclusion Criteria:

* language barrier
* body mass index (BMI) > 40 kg/m2
* multiple gestations
* chronic pain
* opioid use
* substance abuse
* allergies to study medication

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 hours
  24-hour postoperative opioid consumption presented in morphine equivalents

SECONDARY OUTCOMES:
Numeric rating scale pain scores | up to 48 hours
  Pain scores to be assessed at rest and movement 6, 12, 18, 24 and 48 hours post-Cesarean delivery
Time to first analgesia | 48 hours
  Time to request of first analgesia after Cesarean delivery
Opioid side effects | 48 hours
  Evaluate incidence of nausea, vomiting, pruritus, sedation after Cesarean delivery
Patient satisfaction | 48 hours
  Evaluate patient satisfaction of postoperative pain relief at time of discharge
Quality of recovery scores | up to 48 hours
  Quality of recovery (QoR-15) scores acquired preoperatively, 24 hour and 48 hours after Cesarean delivery
Post-discharge numeric rating pain scale scores | up to 60 days
  Evaluate pain scores at 30 days and 60 days after Cesarean delivery

CONTACTS AND LOCATIONS:
Locations (1):
- South Health Campus, Calgary, Alberta, Canada